CLINICAL TRIAL: NCT03898674
Title: Microcirculatory Guided Goal Directed Fluid Therapy in Septic Shock; a Feasibility Study
Acronym: MICRORESUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 40180
Record Dates: First submitted 2019-03-22; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Intervention Model Description: Feasibility study - single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GDT feasibility (Experimental): Patients undergoing microcirculatory goal directed therapy
  Interventions: Drug: Intra venous fluid

INTERVENTIONS:
Drug: Intra venous fluid — Volume of intra venous fluid administered during GDT protocol

SUMMARY:
Prospective single centre study to assess the feasibility of fluid resuscitation guided by macrocirculatory and microcirculation parameters in patients in the early stages of septic shock. The investigators will utilise a novel point of care tool to assess microcirculatory sublingual perfusion in patients with septic shock. This, in combination with conventional haemodynamic monitoring will determine the timing and volume of resuscitative fluid administration. The feasibility of this technique will be determined prior to embarking on a pilot RCT.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years Within 6 hours of ICU admission Evidence of suspected or confirmed infection Serial Organ Failure Assessment (SOFA) score increase of 2 or more (assuming baseline 0 if no previous measures) Requiring vasopressor therapy to maintain a MAP > 65mmHg Lactate > 2 mmol/l despite initial fluid resuscitation Requirement for advanced haemodynamic monitoring (PiCCO system) in the opinion of the attending clinician

Exclusion Criteria:

Patients not expected to survive 24 h in whom the intent of treatment is palliative Patients in whom the primary cause of the shock state is cardiogenic

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-05 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Time to acquire POEM score | 6 hours
  Feasibility measure of point of care test
Effect of POEM score on clinical decision making | 6 hours
  Feasibility outcome measure

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No